CLINICAL TRIAL: NCT03326323
Title: A Pilot Study Involving the Changes in the Markers of Coagulation During Cardiopulmonary Bypass Surgery Utilizing Acute Normovolemic Hemodilution
Brief Title: Biomarker and Thrombogenicity Assessment in Cardiopulmonary Bypass Surgery Utilizing Acute Normovolemic Hemodilution
Acronym: TARGET-ANH
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: Instrumentation Laboratory (Industry)
Responsible Party: Sponsor
Other Study IDs: 172809
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Bleeding Reduction
Keywords: acute normovolemic hemodilution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ANH during CABG: Patients undergoing Acute Normovolemic Hemodilution during CABG surgery.
  Interventions: Procedure: Acute Normovolemic Hemodilution

INTERVENTIONS:
Procedure: Acute Normovolemic Hemodilution — Collection and reinfusion of a patients own blood during coronary artery bypass graft surgery.

SUMMARY:
This study will help enhance current understanding of the impact of Acute Normovolemic Hemodilution (ANH) administration on transfusion requirements post cardiac surgery, the effect of this procedure on coagulation, and platelet hemostasis, and the amount of chest tube drainage 24 hours post coronary artery bypass graft surgery (CABG) surgery.

DETAILED DESCRIPTION:
Acute Normovolemic Hemodilution (ANH) involves the removal of the patients own blood immediately at the induction of anesthesia and replacement of this blood intraoperatively with an equivalent volume of crystalloid or colloid solution in order to dissuade the loss of red blood cell mass, the mechanism of action is dilution of the blood, hematocrit reduction, and reduction of the anticoagulant components of the blood associated with bleeding during cardiopulmonary bypass graft surgery. The collected blood is isolated from the negative effects of the cardiopulmonary bypass machine.. The collected blood is then stored in anticoagulant treated blood bags in the cardiovascular operating room and re-infused into the patient in reverse order of collection at the commencement of surgery, leaving the most cell rich blood to be re-infused into the patient last. This study will evaluate the effect in patients with and without ANH utilization on; hemostatic markers, chest tube drainage 24 hours post CABG, and need for allergenic blood transfusion. Positive effects on the hemostatic markers of anticoagulation and platelets, reduced chest tube drainage at 24 hours post CABG, and reduced number of transfused red blood cells will indicate a positive correlation with ANH utilization during isolated on pump CABG surgery.

The benefits of ANH utilization in blood conservation will benefit patients by reducing their exposure to allogenic blood transfusion with its myriad side effects.

ELIGIBILITY:
Inclusion Criteria:

1. . Subject is 18-85 years old.
2. . Subject is hemodynamically stable
3. . The subject is able to read and has signed and dated the informed consent document including Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization permitting release of personal health information as approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria:

1. . Hematocrit <30 at baseline
2. . Insufficient (Low) on pump hematocrit of < 21%
3. . Patient is hemodynamically unstable
4. . Patient requiring an emergency procedure
5. . Left main coronary artery stenosis with evidence of hemodynamic instability (e.g.. hypotension, ST segment elevations on electrocardiogram)
6. . Aortic valve stenosis with evidence of hemodynamic instability (e.g.. hypotension, ST segment elevations on electrocardiogram)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is inclusive of both genders and all racial and ethnic groups and subgroups. Subjects will be enrolled from age 18-85 years old.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Sarin, MD, Principal Investigator — Inova Heart and Vascular Institute
Locations (1):
- Inova Heart and Vascular Institute, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Undergoing ANH During CABG
Started | 43
Completed | 40
Not Completed | 3
Not completed — Unable to receive ANH protocol | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing ANH During CABG
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Recovery in Platelet Function Post ANH
Description: Time it takes (hours) for platelet function to recover post-ANH to pre-procedure levels as measured by platelet aggregation.
Time Frame: Baseline through 24 hours post ANH procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patients Undergoing ANH During CABG
Number analyzed (Participants) | 40
hours | 2 (30)

2. Secondary Outcome: Recovery in Mean Clot Firmness Post ANH
Description: Time it takes for Mean Clot Firmness (MCF) to return normal levels post-ANH as measured by ROTEM
Time Frame: Baseline through 24 hours post ANH procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patients Undergoing ANH During CABG
Number analyzed (Participants) | 40
hours | 18 (6)

ADVERSE EVENTS:
Time Frame: in-hospital and 30 days
Arm/Group | Patients Undergoing ANH During CABG
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03326323/Prot_SAP_000.pdf